CLINICAL TRIAL: NCT04143594
Title: A Phase 2 Randomized, Open Label, Active Controlled Study Evaluating the Safety and Efficacy of Long-acting Capsid Inhibitor GS-6207 in Combination With Other Antiretroviral Agents in People Living With HIV
Brief Title: Study to Evaluate the Safety and Efficacy of Lenacapavir (GS-6207) in Combination With Other Antiretroviral Agents in People Living With HIV
Acronym: CALIBRATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-200-4334
Record Dates: First submitted 2019-10-28; First posted 2019-10-29 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — lenacapavir; emtricitabine tenofovir alafenamide; imidazole mustard; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lenacapavir, F/TAF, and TAF (Experimental): Induction phase: Participants will receive lenacapavir (LEN) 600 mg (2 X 300 mg, tablet) orally on Days 1 and 2, followed by LEN 300 mg tablet orally on Day 8 plus emtricitabine/ tenofovir alafenamide (F/TAF) (200/25 mg) fixed-dose combination (FDC) tablets once daily orally from Day 1 to Week 28 plus LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via subcutaneous (SC) injection on Day 15.
  Maintenance phase: Participants will receive LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Week 28 and every 6 months (26 weeks) thereafter plus TAF 25 mg tablets once daily orally at Week 28 and will continue up to Week 80.
  Participants willing to continue the study beyond Week 80 will continue to receive SC LEN 927 mg injection every 6 months (26 weeks) and oral daily TAF 25 mg tablets from Week 80 onwards.
  Interventions: Drug: Oral Lenacapavir; Drug: F/TAF; Drug: Subcutaneous Lenacapavir; Drug: TAF
- Lenacapavir, F/TAF, and BIC (Experimental): Induction phase: Participants will receive LEN 600 mg (2 X 300 mg, tablet) orally on Days 1 and 2, followed by LEN 300 mg tablet orally on Day 8 plus F/TAF (200/25 mg) FDC tablets once daily orally from Day 1 to Week 28 plus LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Day 15.
  Maintenance phase: Participants will receive LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Week 28 and every 6 months (26 weeks) thereafter plus bictegravir (BIC) 75 mg tablets once daily orally at Week 28 and will continue up to Week 80.
  Participants willing to continue the study beyond Week 80 will continue to receive SC LEN 927 mg injection every 6 months (26 weeks) and oral daily BIC 75 mg tablets from Week 80 onwards.
  Interventions: Drug: Oral Lenacapavir; Drug: F/TAF; Drug: Subcutaneous Lenacapavir; Drug: BIC
- Lenacapavir and F/TAF (Experimental): Induction phase: Participants will receive LEN 600 mg (2 X 300 mg, tablet) orally on Days 1 and 2, followed by LEN 300 mg tablet orally on Day 8 plus F/TAF (200/25 mg) FDC tablets once daily orally from Day 1 to Week 28 plus LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Day 15.
  Maintenance phase: Participants will receive LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Week 28 and every 6 months (26 weeks) thereafter plus bictegravir (BIC) 75 mg tablets once daily orally at Week 28 and will continue up to Week 80.
  Participants willing to continue the study beyond Week 80 will continue to receive SC LEN 927 mg injection every 6 months (26 weeks) and oral daily BIC 75 mg tablets from Week 80 onwards.
  Interventions: Drug: Oral Lenacapavir; Drug: F/TAF
- B/F/TAF (Active Comparator): Participants will receive bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) FDC tablets once daily orally from Day 1 and throughout their participation in the study up to Week 80
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: Oral Lenacapavir — Tablets administered without regard to food
  Other Names: GS-6207
  Arms: Lenacapavir and F/TAF; Lenacapavir, F/TAF, and BIC; Lenacapavir, F/TAF, and TAF
Drug: F/TAF — Tablets administered without regard to food
  Other Names: Descovy®
  Arms: Lenacapavir and F/TAF; Lenacapavir, F/TAF, and BIC; Lenacapavir, F/TAF, and TAF
Drug: Subcutaneous Lenacapavir — Administered in the abdomen via subcutaneous injections
  Other Names: GS-6207
  Arms: Lenacapavir, F/TAF, and BIC; Lenacapavir, F/TAF, and TAF
Drug: TAF — Tablets administered without regard to food
  Arms: Lenacapavir, F/TAF, and TAF
Drug: BIC — Tablets administered without regard to food
  Arms: Lenacapavir, F/TAF, and BIC
Drug: B/F/TAF — Tablets administered without regard to food
  Other Names: Biktarvy®
  Arms: B/F/TAF

SUMMARY:
The primary objective of this study is to evaluate the efficacy of lenacapavir (formerly GS-6207) containing regimens in people living with human immunodeficiency virus (HIV) (PLWH).

ELIGIBILITY:
Key Inclusion Criteria:

* Antiretroviral (ARV) naive with no use of any ARV within one month of screening. Use of pre-exposure prophylaxis (PrEP) (any duration), post-exposure prophylaxis (PEP) (any duration), or HIV-1 treatment (< 10 days therapy total) > 1 month prior to screening is permitted
* HIV-1 ribonucleic acid (RNA) ≥ 200 copies/mL at screening
* Cluster Determinant 4+ (CD4+) cell count ≥ 200 cells/microliter at screening

Key Exclusion Criteria:

* Current Hepatitis B Virus (HBV) or Hepatitis C virus (HCV) infection

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (53):
- United States (49):
  - Valleywise Community Health Center - McDowell, Phoenix, Arizona
  - Pueblo Family Physicians, Phoenix, Arizona
  - Ruane Clinical Research Group Inc, Los Angeles, California
  - Mills Clinical Research at Men's Health Foundation, Los Angeles, California
  - Eisenhower Health Center at Rimrock, Palm Springs, California
  - University of Colorado, Denver, University of Colorado Hospital, Aurora, Colorado
  - Denver Public Health, Denver, Colorado
  - Yale University; School of Medicine, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Whitman-Walker Institute, Inc., Washington D.C., District of Columbia
  - Washington Health Institute, Washington D.C., District of Columbia
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Floridian Clinical Research, Hialeah, Florida
  - AHF-The Kinder Medical Group, Miami, Florida
  - AIDS Healthcare Foundation - South Beach, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - St. Joseph's Hospital Comprehensive Research Institute, Tampa, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Atlanta ID Group, PC, Atlanta, Georgia
  - August University Medical Center, Augusta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University, Department of Internal Medicine, Macon, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - Howard Brown Health Center, Chicago, Illinois
  - Northstar Healthcare, Chicago, Illinois
  - Indiana University Infectious Diseases Research, Indianapolis, Indiana
  - Be Well Medical Center, Berkley, Michigan
  - St. John Newland Medical Associates, Southfield, Michigan
  - KC CARE Health Center, Kansas City, Missouri
  - AHF-Midtown, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - East Carolina University, The Brody School of Medicine, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Clinical Research Site/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - St Hope Foundation, Bellaire, Texas
  - Prism Health North Texas, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A., Dallas, Texas
  - Texas Centers for Infectious Disease Associates, Fort Worth, Texas
  - The Crofoot Research Center, Inc., Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Clinical Alliance for Research & Education - Infectious Diseases, LLC (CARE-ID), Annandale, Virginia
  - Peter Shalit, M.D., Seattle, Washington
  - MultiCare Rockwood HIV Critical Care Clinic, Spokane, Washington
- Instituto Dominicano de Estudios Virológicos (IDEV), Santo Domingo, Dominican Republic
- Puerto Rico (3):
  - Clinical Research Puerto Rico, San Juan
  - HOPE Clinical Research, San Juan
  - Proyecto ACTU, School of Medicine, University of Puerto Rico, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Background] Gupta SK, Berhe M, Crofoot G, Benson P, Ramgopal M, Sims J, McDonald C, Ruane P, Sanchez WE, Scribner A, Liu SY, VanderVeen LA, Dvory-Sobol H, Rhee MS, Baeten JM, Koenig E. Lenacapavir administered every 26 weeks or daily in combination with oral daily antiretroviral therapy for initial treatment of HIV: a randomised, open-label, active-controlled, phase 2 trial. Lancet HIV. 2023 Jan;10(1):e15-e23. doi: 10.1016/S2352-3018(22)00291-0. PMID 36566079
- [Background] VanderVeen, L. A., et al. Resistance Analysis of Long-Acting Lenacapavir in People With HIV Who are Treatment-Naïve After 80 Weeks of Treatment [Poster14]. European Meeting on HIV & Hepatitis 2023, Rome, Italy.
- [Background] Jogiraju V, Shelton M, Dheri P, Ling J, Wang H, Dvory-Sobol H, et al. Pharmacokinetics of Lenacapavir Alone and When Coadministered With Other Antiretrovirals in People With HIV [Poster PII-056]. American Society for Clinical Pharmacology and Therapeutics (ASCPT) Annual Meeting; 2023 22-24 March; Atlanta, GA.
- [Background] Hagins D, Koenig E, Safran R, Santiago L, Wohlfeiler M, Hsiao C, et al. Long-Acting Lenacapavir in a Combination Regimen for Treatment Naïve PWH: Week 80 [Poster 522]. Conference on Retroviruses and Opportunistic Infections (CROI); 2023 19-22 February; Seattle, WA.
- [Background] VanderVeen LA, Margot N, Naik V, Dvory-Sobol H, Rhee MS, Callebaut C. Resistance Analysis of Long-Acting Lenacapavir in Treatment-Naïve People With HIV at 54 Weeks [Poster EPB239]. AIDS 2022; 2022 29 July-2 August; Montreal, Quebec, Canada.
- [Background] Gupta SK, Sims J, Brinson C, Cruickshank FA, Oguchi G, Morales J, et al. Lenacapavir as part of a Combination Regimen in Treatment-Naïve People with HIV: Week 54 Results [Presentation]. Virtual Conference on Retroviruses and Opportunistic Infections (CROI) 2022; 2022 12-16 February.
- [Background] VanderVeen, L, Margot N, Naik V, et al. Interim Resistance Analysis of Long-Acting Lenacapavir in Treatment-Naïve People with HIV at 28 Weeks (CALIBRATE) [Abstract Oral 73]. Presented at: ID Week; 2021 September 29 - October 03.
- [Background] Gupta SK, Berhe M, Crofoot G, et al. Long-Acting Subcutaneous Lenacapavir Dosed Every 6 Months as part of a Combination Regimen in Treatment-Naïve People with HIV: Interim 16-week Results of a Randomized, Open-label, Phase 2 Induction-Maintenance Study (CALIBRATE) [Abstract OALB0302]. Presented at: International AIDS Society (IAS) Conference; 2021 July 18-21.
- [Derived] Hagins D, Berhe M, Crofoot GE, Ramgopal MN, Sims J, McDonald C, Ruane PJ, Sanchez WE, Scribner A, Benson P, Liu SY, Vanderveen LA, Dvory-Sobol H, Rhee MS, Gupta SK. Final efficacy and safety of twice-yearly subcutaneous lenacapavir in treatment-naive people with HIV: randomized study. AIDS. 2025 Oct 7. doi: 10.1097/QAD.0000000000004372. Online ahead of print. PMID 41056006
- [Derived] Harris P, Henderson R, Hayward P. Highlights from the 11th IAS Conference on Science. Lancet HIV. 2021 Aug;8(8):e459. doi: 10.1016/S2352-3018(21)00161-2. No abstract available. PMID 34358495
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT04143594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Dominican Republic, Puerto Rico, and the United States.
Pre-assignment Details: 249 participants were screened.
Groups:
- Group 1: SC LEN+(F/TAF→ TAF): Induction phase: Participants received lenacapavir (LEN) 600 mg (2 X 300 mg, tablet) orally on Days 1 and 2, followed by LEN 300 mg tablet orally on Day 8 plus emtricitabine/ tenofovir alafenamide (F/TAF) (200/25 mg) fixed-dose combination (FDC) tablets once daily orally from Day 1 to Week 28 plus LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via subcutaneous (SC) injection on Day 15.
  Maintenance phase: Participants received LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Week 28 and every 6 months (26 weeks) thereafter plus TAF 25 mg tablets once daily orally at Week 28 and continued up to Week 80.
  Participants willing to continue the study beyond Week 80 continued to receive SC LEN 927 mg injection every 6 months (26 weeks) and oral daily TAF 25 mg tablets from Week 80 onwards.
- Group 2: SC LEN + (F/TAF → BIC): Induction phase: Participants received LEN 600 mg (2 X 300 mg, tablet) orally on Days 1 and 2, followed by LEN 300 mg tablet orally on Day 8 plus F/TAF (200/25 mg) FDC tablets once daily orally from Day 1 to Week 28 plus LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Day 15.
  Maintenance phase: Participants received LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Week 28 and every 6 months (26 weeks) thereafter plus bictegravir (BIC) 75 mg tablets once daily orally at Week 28 and continued up to Week 80.
  Participants willing to continue the study beyond Week 80 continued to receive SC LEN 927 mg injection every 6 months (26 weeks) and oral daily BIC 75 mg tablets from Week 80 onwards.
- Group 3: Oral LEN + F/TAF: Participants received LEN 600 mg (2 X 300 mg, tablet) orally on Days 1 and 2, followed by LEN 50 mg tablets once daily orally from Day 3 and continued up to Week 80. Participants received F/TAF (200/25 mg) FDC tablets once daily orally from Day 1 and continued up to Week 80.
  Participants willing to continue the study beyond Week 80 continued to receive oral daily LEN 50 mg tablets and oral daily F/TAF 200/25 mg FDC tablets from Week 80 onwards.
- Group 4: B/F/TAF: Participants received bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) FDC tablets once daily orally from Day 1 and throughout their participation in the study up to Week 80.
Period: Overall Study
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Started | 52 | 53 | 52 | 26
Completed | 41 | 35 | 36 | 24
Not Completed | 11 | 18 | 16 | 2
Not completed — Withdrew consent | 3 | 10 | 3 | 1
Not completed — Lost to Follow-up | 3 | 5 | 11 | 0
Not completed — Investigator's discretion | 2 | 2 | 0 | 0
Not completed — Randomized but never treated | 0 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF | Total
Number analyzed (Participants) | 52 | 53 | 52 | 25 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 53 | 51 | 25 | 181
  >=65 years | 0 | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (9.5) | 30 (8.8) | 32 (12.3) | 33 (11.1) | 32 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6 | 0 | 12
  Male | 47 | 52 | 46 | 25 | 170
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Race: Asian | 1 | 0 | 1 | 0 | 2
  Race: Black | 24 | 24 | 31 | 16 | 95
  Race: Native Hawaiian or Pacific Islander | 1 | 1 | 0 | 0 | 2
  Race: White | 23 | 28 | 19 | 8 | 78
  Race: Other | 2 | 0 | 1 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 25 | 21 | 24 | 12 | 82
  Ethnicity: Not Hispanic or Latino | 27 | 32 | 28 | 13 | 100
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 1 | 1 | 5 | 1 | 8
  United States | 37 | 42 | 37 | 21 | 137
  Dominican Republic | 14 | 10 | 10 | 3 | 37
Human Immunodeficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) [Mean (Standard Deviation); unit: log10 copies/mL] | 4.18 (0.672) | 4.35 (0.670) | 4.33 (0.722) | 4.35 (0.780) | 4.30 (0.700)
HIV-1 RNA Categories [Count of Participants; unit: Participants]
  <= 100,000 copies/mL | 47 | 44 | 43 | 21 | 155
  > 100,000 copies/mL | 5 | 9 | 9 | 4 | 27
Clusters of Differentiation 4+ (CD4) Cell Count [Mean (Standard Deviation); unit: cells/μL] | 506 (297.0) | 490 (209.9) | 470 (221.7) | 534 (260.0) | 495 (246.5)
CD4 Cell Count Categories [Count of Participants; unit: Participants]
  < 50 cells/μL | 0 | 0 | 0 | 0 | 0
  >= 50 to < 200 cells/μL | 0 | 1 | 3 | 0 | 4
  >= 200 to < 350 cells/μL | 17 | 15 | 16 | 4 | 52
  >= 350 to < 500 cells/μL | 17 | 15 | 15 | 11 | 58
  >= 500 cells/μL | 18 | 22 | 18 | 10 | 68
CD4 Percentage (%) [Mean (Standard Deviation); unit: percentage of CD4 cells] | 24.2 (9.92) | 24.1 (8.04) | 22.7 (8.28) | 26.2 (8.18) | 24.0 (8.70)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Human Immunodeficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) < 50 Copies/mL at Week 54 as Determined by the United States Food and Drug Administration (US FDA)-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 54 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. Week 54 window was between Day 323 and 413 (inclusive). Percentages were rounded off.
Time Frame: Week 54
Population: Full Analysis Set included all randomized participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Group 1: SC LEN+(F/TAF→ TAF): Induction phase: Participants received lenacapavir (LEN) 600 mg (2 X 300 mg, tablet) orally on Days 1 and 2, followed by LEN 300 mg tablet orally on Day 8 plus emtricitabine/ tenofovir alafenamide (F/TAF) (200/25 mg) fixed-dose combination (FDC) tablets once daily orally from Day 1 to Week 28 plus LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via subcutaneous (SC) injection on Day 15.
  Maintenance phase: Participants received LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Week 28 and every 6 months (26 weeks) thereafter plus TAF 25 mg tablets once daily orally at Week 28 and continued up to Week 80.
  Participants willing to continue the study beyond Week 80 continued to receive SC LEN 927 mg injection every 6 months (26 weeks) and oral daily TAF 25 mg tablets from Week 80 onwards.
  Maintenance phase: Participants received LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Week 28 and every 6 months (26 weeks) thereafter plus TAF 25 mg tablets once daily orally at Week 28 and will continue up to Week 80.
  Participants willing to continue the study beyond Week 80 will continue to receive SC LEN 927 mg injection every 6 months (26 weeks) and oral daily TAF 25 mg tablets from Week 80 onwards.
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 52 | 53 | 52 | 25
percentage of participants | 90.4 | 84.9 | 84.6 | 92.0
Statistical Analysis 1: Comparison: Group 1: SC LEN+(F/TAF→ TAF) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.7178, Cochran-Mantel-Haenszel — P-value was from the Cochran-Mantel-Haenszel (CMH) tests stratified by baseline HIV-1 RNA stratum (≤ 100,000 vs > 100,000 copies/mL); Difference in percentage = -2.6, 95% CI 2-sided [-18.4 to 13.2] — The difference in percentage of participants between LEN-containing and the B/F/TAF groups, and its 95% confidence interval (CI) were calculated based on the MH proportions adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs > 100,000 copies/mL)
Statistical Analysis 2: Comparison: Group 2: SC LEN + (F/TAF → BIC) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.3900, Cochran-Mantel-Haenszel — P-value was from the CMH tests stratified by baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in percentage = -7.1, 95% CI 2-sided [-23.4 to 9.3] — The difference in percentage of participants between LEN-containing treatment groups and the B/F/TAF group, and its 95% CI were calculated based on the MH proportions adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs > 100,000 copies/mL)
Statistical Analysis 3: Comparison: Group 3: Oral LEN + F/TAF vs Group 4: B/F/TAF; Test type: Superiority; p = 0.3797, Cochran-Mantel-Haenszel — P-value was from the CMH tests stratified by baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in percentage = -7.2, 95% CI 2-sided [-23.5 to 9.1] — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 28 as Determined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 28 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. Week 28 window was between Days 176 and 231 (inclusive). Percentages were rounded off.
Time Frame: Week 28
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 52 | 53 | 52 | 25
percentage of participants | 94.2 | 92.5 | 94.2 | 100.0
Statistical Analysis 1: Comparison: Group 1: SC LEN+(F/TAF→ TAF) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.2398, Cochran-Mantel-Haenszel — P-value was from the CMH tests stratified by baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in percentage = -5.5, 95% CI 2-sided [-15.9 to 4.8] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Group 2: SC LEN + (F/TAF → BIC) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.1639, Cochran-Mantel-Haenszel — P-value was from the CMH tests stratified by baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in percentage = -7.4, 95% CI 2-sided [-18.3 to 3.4] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Group 3: Oral LEN + F/TAF vs Group 4: B/F/TAF; Test type: Superiority; p = 0.2307, Cochran-Mantel-Haenszel — P-value was from the CMH tests stratified by baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in percentage = -5.7, 95% CI 2-sided [-16.3 to 4.9] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 38 as Determined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 38 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. Week 38 window was between Days 232 and 322 (inclusive). Percentages were rounded off.
Time Frame: Week 38
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 52 | 53 | 52 | 25
percentage of participants | 90.4 | 88.7 | 88.5 | 96.0
Statistical Analysis 1: Comparison: Group 1: SC LEN+(F/TAF→ TAF) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.3142, Cochran-Mantel-Haenszel — P-value was from the CMH tests stratified by baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in percentage = -6.7, 95% CI 2-sided [-20.7 to 7.3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Group 2: SC LEN + (F/TAF → BIC) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.3009, Cochran-Mantel-Haenszel — P-value was from the CMH tests stratified by baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in percentage = -7.2, 95% CI 2-sided [-21.3 to 6.8] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Group 3: Oral LEN + F/TAF vs Group 4: B/F/TAF; Test type: Superiority; p = 0.2859, Cochran-Mantel-Haenszel — P-value was from the CMH tests stratified by baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in percentage = -7.6, 95% CI 2-sided [-21.8 to 6.7] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 80 as Determined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 80 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status. The Week 80 window was between Days 505 and 595 (inclusive). Percentages were rounded off.
Time Frame: Week 80
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 52 | 53 | 52 | 25
percentage of participants | 86.5 | 75.5 | 86.5 | 92
Statistical Analysis 1: Comparison: Group 1: SC LEN+(F/TAF→ TAF) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.3686, Cochran-Mantel-Haenszel — P-value was from the CMH tests stratified by baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in percentage = -7.1, 95% CI 2-sided [-23.2 to 9.0] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Group 2: SC LEN + (F/TAF → BIC) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.0887, Cochran-Mantel-Haenszel — P-value was from the CMH tests stratified by baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in percentage = -16.5, 95% CI 2-sided [-34.0 to 1.0] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Group 3: Oral LEN + F/TAF vs Group 4: B/F/TAF; Test type: Superiority; p = 0.4949, Cochran-Mantel-Haenszel — P-value was from the CMH tests stratified by baseline HIV-1 RNA stratum (<= 100,000 vs. > 100,000 copies/mL); Difference in percentage = -5.4, 95% CI 2-sided [-21.5 to 10.7] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Change From Baseline in Log10 HIV-1 RNA at Week 28
Time Frame: Baseline, Week 28
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 49 | 51 | 50 | 25
log10 copies/mL | -2.92 (0.649) | -3.04 (0.638) | -3.01 (0.716) | -3.07 (0.774)
Statistical Analysis 1: Comparison: Group 1: SC LEN+(F/TAF→ TAF) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.5755, ANOVA — P-value was from analysis of variance (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 0.08, 95% CI 2-sided [-0.20 to 0.37] — Difference in least squares means (Diff in LSM), and its 95% CI were from ANOVA model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL)
Statistical Analysis 2: Comparison: Group 2: SC LEN + (F/TAF → BIC) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.8697, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 0.02, 95% CI 2-sided [-0.25 to 0.29] — Difference in LSM, and its 95% CI were from ANOVA model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL)
Statistical Analysis 3: Comparison: Group 3: Oral LEN + F/TAF vs Group 4: B/F/TAF; Test type: Superiority; p = 0.7052, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 0.06, 95% CI 2-sided [-0.23 to 0.35] — [estimate comment as in outcome 5, analysis 2]

6. Secondary Outcome: Change From Baseline in Log10 HIV-1 RNA at Week 38
Time Frame: Baseline, Week 38
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 49 | 51 | 47 | 25
log10 copies/mL | -2.96 (0.639) | -3.06 (0.641) | -3.02 (0.771) | -3.04 (0.760)
Statistical Analysis 1: Comparison: Group 1: SC LEN+(F/TAF→ TAF) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.8942, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 0.02, 95% CI 2-sided [-0.26 to 0.30] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Group 2: SC LEN + (F/TAF → BIC) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.9058, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = -0.02, 95% CI 2-sided [-0.28 to 0.25] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Group 3: Oral LEN + F/TAF vs Group 4: B/F/TAF; Test type: Superiority; p = 0.8129, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 0.04, 95% CI 2-sided [-0.27 to 0.35] — [estimate comment as in outcome 5, analysis 2]

7. Secondary Outcome: Change From Baseline in Log10 HIV-1 RNA at Week 54
Time Frame: Baseline, Week 54
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 49 | 47 | 47 | 23
log10 copies/mL | -2.95 (0.636) | -3.12 (0.589) | -2.85 (0.840) | -3.08 (0.787)
Statistical Analysis 1: Comparison: Group 1: SC LEN+(F/TAF→ TAF) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.7864, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 0.04, 95% CI 2-sided [-0.25 to 0.33] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Group 2: SC LEN + (F/TAF → BIC) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.7013, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = -0.05, 95% CI 2-sided [-0.31 to 0.21] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Group 3: Oral LEN + F/TAF vs Group 4: B/F/TAF; Test type: Superiority; p = 0.2753, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 0.22, 95% CI 2-sided [-0.18 to 0.62] — [estimate comment as in outcome 5, analysis 2]

8. Secondary Outcome: Change From Baseline in Log10 HIV-1 RNA at Week 80
Time Frame: Baseline, Week 80
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 Copies/mL
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 48 | 42 | 46 | 24
log10 Copies/mL | -2.96 (0.539) | -3.08 (0.592) | -2.96 (0.747) | -3.09 (0.755)
Statistical Analysis 1: Comparison: Group 1: SC LEN+(F/TAF→ TAF) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.5640, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 0.08, 95% CI 2-sided [-0.19 to 0.34] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Group 2: SC LEN + (F/TAF → BIC) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.9555, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = -0.01, 95% CI 2-sided [-0.28 to 0.26] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Group 3: Oral LEN + F/TAF vs Group 4: B/F/TAF; Test type: Superiority; p = 0.4025, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 0.14, 95% CI 2-sided [-0.19 to 0.46] — [estimate comment as in outcome 5, analysis 2]

9. Secondary Outcome: Change From Baseline in Clusters of Differentiation 4+ (CD4+) Cell Count at Week 28
Time Frame: Baseline, Week 28
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 49 | 50 | 50 | 25
cells/µL | 172 (178.2) | 158 (164.1) | 206 (154.6) | 163 (157.7)
Statistical Analysis 1: Comparison: Group 1: SC LEN+(F/TAF→ TAF) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.7751, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 12, 95% CI 2-sided [-73 to 97] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Group 2: SC LEN + (F/TAF → BIC) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.9549, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = -2, 95% CI 2-sided [-79 to 75] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Group 3: Oral LEN + F/TAF vs Group 4: B/F/TAF; Test type: Superiority; p = 0.2603, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 44, 95% CI 2-sided [-33 to 120] — [estimate comment as in outcome 5, analysis 2]

10. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 38
Time Frame: Baseline, Week 38
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Groups:
- Group 2: SC LEN + (F/TAF → BIC): Induction phase: Participants received lenacapavir (LEN) 600 mg (2 X 300 mg, tablet) orally on Days 1 and 2, followed by LEN 300 mg tablet orally on Day 8 plus emtricitabine/ tenofovir alafenamide (F/TAF) (200/25 mg) fixed-dose combination (FDC) tablets once daily orally from Day 1 to Week 28 plus LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via subcutaneous (SC) injection on Day 15.
  Maintenance phase: Participants received LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Week 28 and every 6 months (26 weeks) thereafter plus TAF 25 mg tablets once daily orally at Week 28 and continued up to Week 80.
  Participants willing to continue the study beyond Week 80 continued to receive SC LEN 927 mg injection every 6 months (26 weeks) and oral daily TAF 25 mg tablets from Week 80 onwards.
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 49 | 51 | 46 | 25
cells/µL | 195 (164.6) | 220 (187.5) | 211 (166.2) | 232 (209.3)
Statistical Analysis 1: Comparison: Group 1: SC LEN+(F/TAF→ TAF) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.4827, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = -31, 95% CI 2-sided [-119 to 57] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Group 2: SC LEN + (F/TAF → BIC) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.7963, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = -12, 95% CI 2-sided [-106 to 81] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Group 3: Oral LEN + F/TAF vs Group 4: B/F/TAF; Test type: Superiority; p = 0.6169, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = -22, 95% CI 2-sided [-111 to 67] — [estimate comment as in outcome 5, analysis 2]

11. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 54
Time Frame: Baseline, Week 54
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 49 | 47 | 47 | 23
cells/µL | 204 (189.1) | 213 (187.2) | 220 (175.5) | 193 (191.1)
Statistical Analysis 1: Comparison: Group 1: SC LEN+(F/TAF→ TAF) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.6614, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 21, 95% CI 2-sided [-73 to 115] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Group 2: SC LEN + (F/TAF → BIC) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.6791, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 20, 95% CI 2-sided [-75 to 115] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Group 3: Oral LEN + F/TAF vs Group 4: B/F/TAF; Test type: Superiority; p = 0.5563, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 27, 95% CI 2-sided [-65 to 120] — [estimate comment as in outcome 5, analysis 2]

12. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 80
Time Frame: Baseline, Week 80
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 48 | 41 | 46 | 24
cells/μL | 275 (211.8) | 262 (184.4) | 245 (237.4) | 248 (218.7)
Statistical Analysis 1: Comparison: Group 1: SC LEN+(F/TAF→ TAF) vs Group 4: B/F/TAF; Test type: Superiority; p = 0.5492, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 32, 95% CI 2-sided [-75 to 140] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Group 2: SC LEN + (F/TAF → BIC); Test type: Superiority; p = 0.7220, Difference in LSM — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = 17, 95% CI 2-sided [-80 to 115] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Group 3: Oral LEN + F/TAF vs Group 4: B/F/TAF; Test type: Superiority; p = 0.9486, ANOVA — P-value was from (ANOVA) model adjusting for the baseline HIV-1 RNA level (<= 100,000 copies/mL or > 100,000 copies/mL); Difference in LSM = -4, 95% CI 2-sided [-118 to 110] — [estimate comment as in outcome 5, analysis 2]

13. Secondary Outcome: Percentage of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as 1 or both of any AEs leading to premature discontinuation of study drug, or any AEs with an onset date on or after the study drug start date and no later than the last exposure date after permanent discontinuation of the study drug. Percentages were rounded off.
Time Frame: Up to 174.9 weeks
Population: Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 52 | 53 | 52 | 25
percentage of participants | 98.1 | 88.7 | 90.4 | 84.0

14. Secondary Outcome: Percentage of Participants Who Experienced Maximum Postbaseline Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least 1 toxicity grade from baseline at any postbaseline visit, up to last exposure date for participants who permanently discontinued study drug. Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening. Percentages were rounded off.
Time Frame: Up to 174.9 weeks
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
Number analyzed (Participants) | 52 | 53 | 52 | 25
percentage of participants
  Grade 1 | 9.6 | 3.8 | 9.6 | 0
  Grade 2 | 55.8 | 56.6 | 42.3 | 76.0
  Grade 3 | 17.3 | 28.3 | 30.8 | 24.0
  Grade 4 | 13.5 | 9.4 | 13.5 | 0

15. Secondary Outcome: Pharmacokinetics (PK) of LEN: Plasma LEN Pre-dose Concentrations for SC LEN
Time Frame: Day 2, 8, Day 1 SC (Day 15), Week 28 and Week 54
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC)
Number analyzed (Participants) | 52 | 53
ng/mL
  Day 2: number analyzed (Participants) | 52 | 52
  Day 2 | 28.3 (27.15) | 26.1 (20.46)
  Day 8: number analyzed (Participants) | 52 | 52
  Day 8 | 34.5 (20.96) | 32.1 (14.71)
  Day 1 SC (Day 15): number analyzed (Participants) | 51 | 52
  Day 1 SC (Day 15) | 30.9 (16.76) | 31.2 (14.66)
  Week 28: number analyzed (Participants) | 49 | 47
  Week 28 | 22.0 (11.70) | 23.0 (14.81)
  Week 54: number analyzed (Participants) | 49 | 43
  Week 54 | 26.9 (14.19) | 26.4 (12.10)

16. Secondary Outcome: PK of LEN : Plasma LEN Single Anytime Concentrations for the Oral LEN + DVY
Time Frame: Day 2, 8, 15 , Week 28 and Week 54
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 3: Oral LEN + F/TAF
Number analyzed (Participants) | 52
ng/mL
  Day 2 | 29.8 (42.70)
  Day 8: number analyzed (Participants) | 50
  Day 8 | 78.7 (55.90)
  Day 15: number analyzed (Participants) | 49
  Day 15 | 97.2 (67.25)
  Week 28: number analyzed (Participants) | 49
  Week 28 | 96.6 (76.40)
  Week 54: number analyzed (Participants) | 46
  Week 54 | 98.4 (85.25)

17. Secondary Outcome: PK of TAF (Tenofovir Alafenamide) and TFV (Tenofovir): Area Under the Concentration Versus Time Curve (AUClast) on Day 1
Description: AUClast is defined as area under the concentration versus time curve from time zero to the last quantifiable concentration. A PK substudy was conducted in at least 10 participants in each of the treatment groups receiving SC LEN (Treatment Groups 1 and 2) and at least 15 participants in the treatment group receiving oral LEN (Treatment Group 3). Key PK parameters of TAF and TFV were summarized for participants in the PK Sub study Analysis Set by treatment group, analyte and visit. PK substudy analysis was conducted for Group 1 and 2 on Day 1.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose on Day 1
Population: PK Substudy Analysis Set included participants who were randomized into the study, were enrolled into the PK Substudy, had received at least 1 dose of active study drug, and had at least 1 nonmissing intensive PK substudy concentration value for any analyte of interest reported by the PK lab.
Measure: Mean (Standard Deviation); unit: hours*nanogram/mL (h*ng/mL)
Groups:
- Group 1: SC LEN+(F/TAF→ TAF): Induction phase: Participants received LEN 600 mg (2 X 300 mg, tablet) orally on Days 1 and 2, followed by LEN 300 mg tablet orally on Day 8 plus F/TAF (200/25 mg) FDC tablets once daily orally from Day 1 to Week 28 plus LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Day 15.
  Maintenance phase: Participants received LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Week 28 and every 6 months (26 weeks) thereafter plus TAF 25 mg tablets once daily orally at Week 28 and will continue up to Week 80.
  Participants willing to continue the study beyond Week 80 will continue to receive SC LEN 927 mg injection every 6 months (26 weeks) and oral daily TAF 25 mg tablets from Week 80 onwards.
- Group 2: SC LEN + (F/TAF → BIC): Induction phase: Participants received LEN 600 mg (2 X 300 mg, tablet) orally on Days 1 and 2, followed by LEN 300 mg tablet orally on Day 8 plus F/TAF (200/25 mg) FDC tablets once daily orally from Day 1 to Week 28 plus LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Day 15.
  Maintenance phase: Participants received LEN 927 mg (309 mg/mL; 2 X 1.5 mL) via SC injection on Week 28 and every 6 months (26 weeks) thereafter plus BIC 75 mg tablets once daily orally at Week 28 and will continue up to Week 80.
  Participants willing to continue the study beyond Week 80 will continue to receive SC LEN 927 mg injection every 6 months (26 weeks) and oral daily BIC 75 mg tablets from Week 80 onwards.
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC)
Number analyzed (Participants) | 10 | 14
hours*nanogram/mL (h*ng/mL)
  TAF | 298.0 (88.0) | 260.0 (63.5)
  TFV: number analyzed (Participants) | 4 | 9
  TFV | 27.1 (27.9) | 40.5 (59.7)

18. Secondary Outcome: PK of TAF and TFV (Tenofovir): Maximum Observed Concentration of Drug (Cmax) on Day 1
Description: Cmax is defined as the maximum observed concentration of drug. A PK substudy was conducted in at least 10 participants in each of the treatment groups receiving SC LEN (Treatment Groups 1 and 2). Key PK parameters of TAF and TFV were summarized for participants in the PK Sub study Analysis Set by treatment group, analyte and visit. PK substudy analysis was conducted for Group 1 and 2 on Day 1.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose on Day 1
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC)
Number analyzed (Participants) | 10 | 14
ng/mL
  TAF | 278.8 (87.7) | 318.4 (57.7)
  TFV: number analyzed (Participants) | 4 | 9
  TFV | 5.4 (26.5) | 13.8 (160.2)

19. Secondary Outcome: PK of TAF and TFV: Time (Observed Time Point) of Cmax (Tmax) on Day 1
Description: Tmax is defined as the time (observed time point) of Cmax. A PK substudy was conducted in at least 10 participants in each of the treatment groups receiving SC LEN (Treatment Groups 1 and 2). Key PK parameters of TAF and TFV were summarized for participants in the PK Sub study Analysis Set by treatment group, analyte and visit. PK substudy analysis was conducted for Group 1 and 2 on Day 1.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose on Day 1
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC)
Number analyzed (Participants) | 10 | 14
hours
  TAF | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 0.50]
  TFV: number analyzed (Participants) | 4 | 9
  TFV | 1.50 [1.00 to 2.02] | 1.00 [0.50 to 1.17]

20. Secondary Outcome: PK of TFV: Last Observed Quantifiable Concentration of the Drug (Clast) on Day 1
Description: Clast is defined as the last observable concentration of drug. A PK substudy was conducted in at least 10 participants in each of the treatment groups receiving SC LEN (Treatment Groups 1 and 2). Key PK parameters of TFV were summarized for participants in the PK Sub study Analysis Set by treatment group, analyte and visit. PK sub study analysis was conducted for Group 1 and 2 on Day 1.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose on Day 1
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC)
Number analyzed (Participants) | 4 | 9
ng/mL | 2.7 (23.1) | 3.9 (38.0)

21. Secondary Outcome: PK of TAF and TFV: AUClast at Weeks 16, 22, or 28
Description: AUClast is defined as area under the concentration versus time curve from time zero to the last quantifiable concentration. A PK substudy was conducted in at least 15 participants in the treatment group receiving oral LEN (Treatment Group 3). Key PK parameters of TAF and TFV were summarized for participants in the PK Sub study Analysis Set by treatment group, analyte and visit. For each participant, PK samples were taken at only one of the three possible visits: Weeks 16, 22, or 28. The PK results were combined and summarized without regard to specific study visit within the range of prespecified study visits.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group 3: Oral LEN + F/TAF
Number analyzed (Participants) | 12
h*ng/mL
  TAF | 231.2 (60.0)
  TFV | 173.1 (52.5)

22. Secondary Outcome: PK of TAF and TFV: Cmax at Weeks 16, 22, or 28
Description: Cmax is defined as the maximum observed concentration of drug. A PK substudy was conducted in at least 15 participants in the treatment group receiving oral LEN (Treatment Group 3). Key PK parameters of TAF and TFV were summarized for participants in the PK Sub study Analysis Set by treatment group, analyte and visit. For each participant, PK samples were taken at only one of the three possible visits: Weeks 16, 22, or 28. The PK results were combined and summarized without regard to specific study visit within the range of prespecified study visits.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 3: Oral LEN + F/TAF
Number analyzed (Participants) | 12
ng/mL
  TAF | 308.7 (74.7)
  TFV | 31.2 (51.7)

23. Secondary Outcome: PK of TAF and TFV: Tmax at Weeks 16, 22, or 28
Description: Tmax is defined as the time (observed time point) of Cmax. A PK substudy was conducted in at least 15 participants in the treatment group receiving oral LEN (Treatment Group 3). Key PK parameters of TAF and TFV were summarized for participants in the PK Sub study Analysis Set by treatment group, analyte and visit. For each participant, PK samples were taken at only one of the three possible visits: Weeks 16, 22, or 28. The PK results were combined and summarized without regard to specific study visit within the range of prespecified study visits.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Group 3: Oral LEN + F/TAF
Number analyzed (Participants) | 12
hours
  TAF | 0.53 [0.50 to 1.04]
  TFV | 1.00 [1.00 to 2.00]

24. Secondary Outcome: PK of TFV: Clast at Weeks 16, 22, or 28
Description: Clast is defined as the last observable concentration of drug. A PK substudy was conducted in at least 15 participants in the treatment group receiving oral LEN (Treatment Group 3). Key PK parameters of TFV was summarized for participants in the PK Sub study Analysis Set by treatment group, analyte and visit. For each participant, PK samples were taken at only one of the three possible visits: Weeks 16, 22, or 28. The PK results were combined and summarized without regard to specific study visit within the range of prespecified study visits.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 3: Oral LEN + F/TAF
Number analyzed (Participants) | 12
ng/mL | 22.2 (62.6)

25. Secondary Outcome: PK of TAF: AUClast at Week 38
Description: AUClast is defined as area under the concentration versus time curve from time zero to the last quantifiable concentration. A PK substudy was conducted in at least 10 participants in each of the treatment groups receiving SC LEN (Treatment Groups 1 and 2). Key PK parameters of TAF was summarized for participants in the PK Sub study Analysis Set by treatment group, analyte and visit. PK substudy analysis was conducted for Group 1 at Week 38.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF)
Number analyzed (Participants) | 11
h*ng/mL | 211.5 (74.1)

26. Secondary Outcome: PK of TAF: Cmax at Week 38
Description: Cmax is defined as the maximum observed concentration of drug. A PK substudy was conducted in at least 10 participants in each of the treatment groups receiving SC LEN (Treatment Groups 1 and 2). Key PK parameters of TAF was summarized for participants in the PK Sub study Analysis Set by treatment group, analyte and visit. PK substudy analysis was conducted for Group 1 at Week 38.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF)
Number analyzed (Participants) | 11
ng/mL | 279.0 (67.8)

27. Secondary Outcome: PK of TAF: Tmax at Week 38
Description: Tmax is defined as the time (observed time point) of Cmax. A PK substudy was conducted in at least 10 participants in each of the treatment groups receiving SC LEN (Treatment Groups 1 and 2). Key PK parameters of TAF was summarized for participants in the PK Sub study Analysis Set by treatment group, analyte and visit. PK substudy analysis was conducted for Group 1 at Week 38.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF)
Number analyzed (Participants) | 11
hours | 0.50 [0.50 to 0.50]

28. Secondary Outcome: PK of Tenofovir Diphosphate (TFV-DP): AUClast at Weeks 4, 10, 16, or 22
Description: AUClast is defined as area under the concentration versus time curve from time zero to the last quantifiable concentration. A peripheral blood mononuclear cell (PBMC) substudy was conducted in a total of approximately 15 participants in Treatment Groups 1 and 2. For each participant, PK samples were taken at only one of the four possible visits: Weeks 4, 10, 16, or 22. A 12-hour postdose sample was collected, if possible. The PK results were combined and summarized without regard to specific study visit within the range of prespecified study visits.
Time Frame: 0 hours (Predose) and at 1, 2, and 6 hours postdose
Population: The PBMC PK Substudy Analysis Set included all randomized participants who took at least 1 dose of study drug, participated in the PBMC substudy, and have at least 1 nonmissing postdose concentration value for tenofovir diphosphate (TFV-DP). The PBMC PK Substudy Analysis Set was used for PK analyses of TFV-DP.
Measure: Mean (Standard Deviation); unit: h*μM
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC)
Number analyzed (Participants) | 13 | 13
h*μM | 16.2 (68.3) | 21.6 (71.9)

29. Secondary Outcome: PK of TFV-DP: Cmax at Weeks 4, 10, 16, or 22
Description: Cmax is defined as the maximum observed concentration of drug. A PBMC substudy was conducted in a total of approximately 15 participants in Treatment Groups 1 and 2. For each participant, PK samples were taken at only one of the four possible visits: Weeks 4, 10, 16, or 22. A 12-hour postdose sample was collected, if possible. The PK results were combined and summarized without regard to specific study visit within the range of prespecified study visits.
Time Frame: 0 hours (Predose) and at 1, 2, and 6 hours postdose
Population: Participants in the PBMC PK Substudy Analysis Set with the available data were analyzed.
Measure: Mean (Standard Deviation); unit: micrometer (μM)
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC)
Number analyzed (Participants) | 13 | 13
micrometer (μM) | 3.3 (37.5) | 4.3 (71.8)

30. Secondary Outcome: PK of TFV-DP: Tmax at Weeks 4, 10, 16, or 22
Description: Tmax is defined as the time (observed time point) of Cmax. A PBMC substudy was conducted in a total of approximately 15 participants in Treatment Groups 1 and 2. For each participant, PK samples were taken at only one of the four possible visits: Weeks 4, 10, 16, or 22. A 12-hour postdose sample was collected, if possible. The PK results were combined and summarized without regard to specific study visit within the range of prespecified study visits.
Time Frame: 0 hours (Predose) and at 1, 2, and 6 hours postdose
Population: Participants in the PBMC PK Substudy Analysis Set with the available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC)
Number analyzed (Participants) | 13 | 13
hours | 2.00 [1.00 to 6.00] | 6.00 [1.00 to 6.00]

31. Secondary Outcome: PK of Bictegravir (BIC): AUClast at Week 38
Description: AUClast is defined as area under the concentration versus time curve from time zero to the last quantifiable concentration. A PK substudy was conducted in at least 10 participants in each of the treatment groups receiving SC LEN (Treatment Groups 1 and 2). At Week 38, samples were analyzed for BIC only in Treatment Group 2.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group 2: SC LEN + (F/TAF → BIC)
Number analyzed (Participants) | 11
h*ng/mL | 72865.9 (31.0)

32. Secondary Outcome: PK of BIC: Cmax at Week 38
Description: Cmax is defined as the maximum observed concentration of drug. A PK substudy was conducted in at least 10 participants in each of the treatment groups receiving SC LEN (Treatment Groups 1 and 2). At Week 38, samples were analyzed for BIC only in Treatment Group 2.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 2: SC LEN + (F/TAF → BIC)
Number analyzed (Participants) | 12
ng/mL | 10180.0 (42.8)

33. Secondary Outcome: PK of BIC: Tmax at Week 38
Description: Tmax is defined as the time (observed time point) of Cmax. A PK substudy was conducted in at least 10 participants in each of the treatment groups receiving SC LEN (Treatment Groups 1 and 2). At Week 38, samples were analyzed for BIC only in Treatment Group 2.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Group 2: SC LEN + (F/TAF → BIC)
Number analyzed (Participants) | 12
hours | 2.00 [1.00 to 3.00]

34. Secondary Outcome: PK of BIC: Clast at Week 38
Description: Clast is defined as the last observable concentration of drug. A PK substudy was conducted in at least 10 participants in each of the treatment groups receiving SC LEN (Treatment Groups 1 and 2). At Week 38, samples were analyzed for BIC only in Treatment Group 2.
Time Frame: 0 hours (Predose) and at 0.5, 1, 2, 3, 4, 5, 6, and 8 hours postdose
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 2: SC LEN + (F/TAF → BIC)
Number analyzed (Participants) | 12
ng/mL | 8474.5 (33.3)

ADVERSE EVENTS:
Time Frame: Adverse Events: Up to 174.9 weeks ; All-Cause Mortality: Up to 189 weeks
Description: All-cause mortality: All Randomized Analysis Set included all participants who were randomized in the study.
  Adverse events: Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Group 3: Oral LEN + F/TAF: Participants received LEN 600 mg (2 X 300 mg, tablet) orally on Days 1 and 2, followed by LEN 50 mg tablets once daily orally from Day 3 and will continue up to Week 80. Participants received F/TAF (200/25 mg) FDC tablets once daily orally from Day 1 and will continue up to Week 80.
  Participants willing to continue the study beyond Week 80 will continue to receive oral daily LEN 50 mg tablets and oral daily F/TAF 200/25 mg FDC tablets from Week 80 onwards.
- Group 4: B/F/TAF: Participants received B/F/TAF (50/200/25 mg) FDC tablets once daily orally from Day 1 and throughout their participation in the study up to Week 80.
Arm/Group | Group 1: SC LEN+(F/TAF→ TAF) | Group 2: SC LEN + (F/TAF → BIC) | Group 3: Oral LEN + F/TAF | Group 4: B/F/TAF
All-Cause Mortality (participants affected / at risk) | 1/52 | 0/53 | 1/52 | 0/26
Serious Adverse Events (participants affected / at risk) | 4/52 | 4/53 | 7/52 | 0/25
Other Adverse Events (participants affected / at risk) | 47/52 | 46/53 | 42/52 | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: SC LEN+(F/TAF→ TAF) (N=52) | Group 2: SC LEN + (F/TAF → BIC) (N=53) | Group 3: Oral LEN + F/TAF (N=52) | Group 4: B/F/TAF (N=25)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Loss of personal independence in daily activities (Social circumstances) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: SC LEN+(F/TAF→ TAF) (N=52) | Group 2: SC LEN + (F/TAF → BIC) (N=53) | Group 3: Oral LEN + F/TAF (N=52) | Group 4: B/F/TAF (N=25)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 | 4 | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 8 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 3 | 1 | 2
Nausea (Gastrointestinal disorders) | 10 | 5 | 7 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1 | 6 | 0
Fatigue (General disorders) | 2 | 7 | 3 | 1
Injection site erythema (General disorders) | 25 | 18 | 0 | 0
Injection site induration (General disorders) | 11 | 11 | 0 | 0
Injection site inflammation (General disorders) | 12 | 4 | 0 | 0
Injection site nodule (General disorders) | 11 | 13 | 0 | 0
Injection site pain (General disorders) | 15 | 14 | 0 | 0
Injection site swelling (General disorders) | 17 | 18 | 0 | 0
Pyrexia (General disorders) | 4 | 2 | 3 | 1
Hypersensitivity (Immune system disorders) | 2 | 3 | 1 | 1
Acarodermatitis (Infections and infestations) | 3 | 0 | 1 | 1
Anal chlamydia infection (Infections and infestations) | 0 | 2 | 5 | 0
Anal gonococcal infection (Infections and infestations) | 0 | 2 | 3 | 0
Body tinea (Infections and infestations) | 3 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 10 | 9 | 11 | 4
Gonorrhoea (Infections and infestations) | 3 | 4 | 5 | 1
Influenza (Infections and infestations) | 13 | 5 | 11 | 0
Nasopharyngitis (Infections and infestations) | 9 | 6 | 5 | 0
Onychomycosis (Infections and infestations) | 4 | 2 | 2 | 0
Oropharyngeal gonococcal infection (Infections and infestations) | 3 | 1 | 5 | 1
Otitis media (Infections and infestations) | 2 | 1 | 1 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 3 | 1 | 0
Secondary syphilis (Infections and infestations) | 2 | 3 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 4 | 1 | 0
Syphilis (Infections and infestations) | 8 | 9 | 7 | 4
Tinea versicolour (Infections and infestations) | 3 | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 3 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 1 | 7 | 3
Urinary tract infection (Infections and infestations) | 1 | 2 | 4 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 4 | 3 | 3 | 1
Weight increased (Investigations) | 3 | 4 | 2 | 3
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 3 | 3 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 4 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 2
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 1
Dizziness (Nervous system disorders) | 4 | 2 | 2 | 1
Headache (Nervous system disorders) | 10 | 8 | 9 | 3
Anxiety (Psychiatric disorders) | 3 | 3 | 4 | 2
Depression (Psychiatric disorders) | 2 | 6 | 4 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 3
Proteinuria (Renal and urinary disorders) | 3 | 1 | 6 | 1
Testicular pain (Reproductive system and breast disorders) | 2 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 5 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 4 | 1
Hypertension (Vascular disorders) | 4 | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT04143594/Prot_000.pdf
  • Statistical Analysis Plan: Week 28 Analysis (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04143594/SAP_001.pdf
  • Statistical Analysis Plan: Week 54 Analysis (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT04143594/SAP_002.pdf
  • Statistical Analysis Plan: Week 80 Final Analysis (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT04143594/SAP_003.pdf